CLINICAL TRIAL: NCT04685174
Title: Intraoperative Near Infrared Spectroscopy of Transplanted Kidney for Prediction of Acute and Sub-acute Kidney Injury in Transplanted Patients
Brief Title: Intraoperative NIRS of Transplanted Kidney for Prediction of Acute and Sub-acute Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-20-OG-0143-20-CTIL
Record Dates: First submitted 2020-11-09; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Graft Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Invos Model 5100C Cerebral/Somatic Oximeter — To measure the correlation between post arterial and venous anastomoses (reperfusion) NIRS values of transplanted kidney and post-transplant graft failure as manifested in initiation of renal replacement therapy post transplant

SUMMARY:
This is a prospective, observational cohort study, designed to explore the use of NIRS in kidney transplants. This study will investigate an association between measurements of intra- operative NIRS and post - operative graft dysfunction as manifested in initiation of renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidates (living/ cadaver donor) at TLVMC who will consent to participate.

Exclusion Criteria:

* Patients unable to give consent,
* patients whose surgeries were aborted before transplant,
* patients who were lost to follow up during the first 7 post-transplant days,
* patients who suffered from surgical graft failure (vascular problems or need for re exploration due to bleeding etc.)
* No pregnant patients will participate in this study.
* No minors will participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Graft Failure | 7 days post operative
  Initiation of renal replacement therapy
Graft Failure | 6 months post operative
  Initiation of renal replacement therapy

IPD SHARING:
Plan to Share IPD: No